CLINICAL TRIAL: NCT01835223
Title: Multicenter Phase 1b/2 Study of Tivozanib in Patients With Advanced Inoperable Hepatocellular Carcinoma
Brief Title: Tivozanib in Treating Patients With Liver Cancer That Is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); AVEO Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I 229112; NCI-2013-00756 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 229112 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Advanced Adult Hepatocellular Carcinoma; Non-Resectable Hepatocellular Carcinoma
MeSH Terms: interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (tivozanib - 1 mg) (Experimental): Patients receive tivozanib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tivozanib (1mg)
- Treatment (tivozanib - 1.5 mg) (Experimental): Patients receive tivozanib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tivozanib (1.5mg)

INTERVENTIONS:
Drug: Tivozanib (1mg) — Given PO
  Other Names: AV-951; TIVOZANIB
  Arms: Treatment (tivozanib - 1 mg)
Drug: Tivozanib (1.5mg) — Given PO
  Other Names: AV-951; TIVOZANIB
  Arms: Treatment (tivozanib - 1.5 mg)

SUMMARY:
This phase I/II trial studies the side effects and best dose of tivozanib and to see how well it works in treating patients with liver cancer that has spread to other parts of the body or cannot be removed by surgery. Tivozanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Progression free survival (PFS) at 24 weeks in patients with advanced hepatocellular carcinoma (HCC).

SECONDARY OBJECTIVES:

I. To determine the safety of tivozanib in HCC. II. To determine the overall survival (OS) and clinical benefit rate (complete response [CR], partial response [PR] and stable disease [SD]) by Response Evaluation Criteria in Solid Tumors (RECIST).

III. To determine the steady state pharmacokinetics (PK) and soluble vascular endothelial growth factor receptor 2 (VEGFR-2) baseline/change with tivozanib and use modeling to correlate exposure with biomarker change and the primary outcome measure of PFS.

IV. To determine the change in viral load (hepatitis B virus [HBV] and hepatitis C virus [HCV]) during therapy in patients with HBV or HCV associated HCC.

V. To determine the change in tumor marker (alfa fetoprotein) with tivozanib therapy is in the effect of tivozanib on several tumor-associated immune response markers.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive tivozanib orally (PO) once daily (QD) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced staged HCC (unresectable and not amenable to local or regional therapy; or metastatic HCC); the diagnosis of HCC should be based on at least one of the following:

  * Magnetic resonance imaging (MRI) or computed tomography (CT) consistent with liver cirrhosis AND at least one solid liver lesion measuring >= 2 cm, with characteristics arterial enhancement and venous washout regardless of alpha-fetoprotein (AFP) levels
  * AFP >= 400 ng/mL AND evidence of at least one solid liver lesion >= 2 cm regardless of specific imaging characteristics on CT or MRI
  * Histological/cytology biopsy confirming HCC
* Patients must have measurable disease per RECIST 1.1 criteria defined as at least one lesion that can be accurately measured in at least one dimension, and that has not been the target of local or regional therapy including transarterial chemoembolization, intra-arterial chemotherapy, ethanol or radiofrequency ablation
* Life expectancy of greater than 3 months
* Child-Pugh liver function class A
* Aspartate aminotransferase (AST) =< 5 x institutional upper limits of normal (ULN)
* Total bilirubin =< 3 mg/dL
* International normalized ratio (INR) =< 2.0 (unless due to therapeutic warfarin use)
* Serum albumin > 2.8 g/dL
* Creatinine =< 1.5 x institutional ULN
* Absolute neutrophil count (ANC) >= 1200/mm^3
* Platelets >= 60,000/mm^3
* Hemoglobin (Hgb) >= 8.5 g/dL
* Patients must not have any evidence of bleeding diathesis or active gastrointestinal bleeding
* Patients must not be known to be human immunodeficiency virus (HIV) positive
* Patients must not have other uncontrolled intercurrent illnesses (excluding HBV or HCV); this includes (but is not limited to) ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Sexually active fertile patients (male and female), and their partners, must agree to use medically accepted methods of contraception during the course of the study and for 3 months after the last dose of the study drug
* Female patients of childbearing potential must have a negative pregnancy test at screening
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients who have had prior anti-angiogenic therapy, including but not limited to sorafenib, brivanib, bevacizumab, or sunitinib
* Patients who have had any prior line of systemic therapy including cytotoxic agents or molecularly targeted agents for advanced/unresectable disease; any number of prior regional therapies with transarterial chemoembolization (TACE), brachytherapy with yttrium-90 microsphere, intra-arterial chemotherapy, surgery, or ablative therapy are allowed
* Prior liver transplantation and on immunosuppression
* Known symptomatic or uncontrolled brain metastases or epidural disease
* Patient has a corrected QT interval (QTcF) > 500 ms at screening
* The patient is unable to swallow pills or diagnosed with a gastrointestinal disorder that are likely to interfere with the absorption of the study drug or with the patient's ability to take regular oral medication
* The patient is pregnant or breastfeeding
* Patients with second primary cancer (except adequately treated nonmelanoma skin cancer, curatively treated in-situ carcinoma of the cervix or superficial bladder cancer, or other solid tumors including lymphoma without bone marrow involvement curatively treated with no evidence of disease for >= 5 years)
* The patient has a previously-identified allergy or hypersensitivity to components of the study treatment formulation
* Patients receiving any medications or substances that are strong inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible; moderate inducers of CYP3A4 should be used with caution
* Urine protein: creatinine ratio > 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Derived] Kalathil SG, Thanavala Y. Natural Killer Cells and T Cells in Hepatocellular Carcinoma and Viral Hepatitis: Current Status and Perspectives for Future Immunotherapeutic Approaches. Cells. 2021 May 28;10(6):1332. doi: 10.3390/cells10061332. PMID 34071188
- [Derived] Kalathil SG, Thanavala Y. Importance of myeloid derived suppressor cells in cancer from a biomarker perspective. Cell Immunol. 2021 Mar;361:104280. doi: 10.1016/j.cellimm.2020.104280. Epub 2020 Dec 31. PMID 33445053
- [Derived] Kalathil SG, Wang K, Hutson A, Iyer R, Thanavala Y. Tivozanib mediated inhibition of c-Kit/SCF signaling on Tregs and MDSCs and reversal of tumor induced immune suppression correlates with survival of HCC patients. Oncoimmunology. 2020 Sep 30;9(1):1824863. doi: 10.1080/2162402X.2020.1824863. PMID 33101775
- [Derived] Fountzilas C, Gupta M, Lee S, Krishnamurthi S, Estfan B, Wang K, Attwood K, Wilton J, Bies R, Bshara W, Iyer R. A multicentre phase 1b/2 study of tivozanib in patients with advanced inoperable hepatocellular carcinoma. Br J Cancer. 2020 Mar;122(7):963-970. doi: 10.1038/s41416-020-0737-6. Epub 2020 Feb 10. PMID 32037403

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Tivozanib 1mg): Patients receive tivozanib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Tivozanib: Given PO
- Treatment (Tivozanib 1.5mg): Patients receive tivozanib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Started | 30 | 3
Completed | 21 | 2
Not Completed | 9 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Disease progression | 2 | 1
Not completed — Became Inelligible | 4 | 0

BASELINE CHARACTERISTICS:
Population: Only 27 patient received any treatment.
Groups:
- Treatment (Tivozanib 1.5mg): Patients receive tivozanib PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Tivozanib: Given PO
- Total: Total of all reporting groups
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg) | Total
Number analyzed (Participants) | 24 | 3 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 1 | 10
  >=65 years | 15 | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (5.5) | 65.5 (11.4) | 65.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 23 | 3 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 22 | 3 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 3 | 27
ECOG Performance Status [Number; unit: participants] — ECOG 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  participants
    0:Fully active, able to carry on all pre-disease performance without restriction. | 14 | 2 | 16
    1: Restricted in physically strenuous, but able for work of light or sedentary nature | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: PFS, Assessed Using Standard RECIST Criteria
Description: Will be descriptively analyzed using standard Kaplan-Meier estimation along with the corresponding descriptive statistics and 95% confidence intervals.
Time Frame: 24 weeks
Population: This outcome was only assessed as part of the Phase II study - which was conducted on the Tivozanib 1mg arm.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Number analyzed (Participants) | 19 | 0
percentage of participants | 58 [33 to 76] |

2. Secondary Outcome: Clinical Benefit Rate (CR, PR, and SD) by RECIST
Description: The number of patients achieving clinical benefit (CR, PR, or SD by RECIST).
Time Frame: Up to 3 years
Population: This outcome was only assessed as part of the Phase II study - which was conducted on the Tivozanib 1mg arm.
  Only 19 subjects were evaluable for the primary or secondary end-points.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib - 1 mg) | Treatment (Tivozanib - 1.5 mg)
Number analyzed (Participants) | 19 | 0
Participants | 12 |

3. Secondary Outcome: Incidence of Adverse Events and Toxicities, Assessed Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4
Description: Toxicity frequency will be tabulated by grade across all dose levels and cycles for all patients in the safety sample and for the subset treated at the recommended phase 2 dose.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Number analyzed (Participants) | 19 | 0
Participants | 19 |

4. Secondary Outcome: Overall Survival Rate
Description: Overall survival is defined as the time from treatment until death or last follow-up.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percent probability
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Number analyzed (Participants) | 19 | 0
percent probability | 0.40 [0.19 to 0.60] |

5. Other Pre Specified Outcome: AFP Response
Description: Defined as an AFP decrease greater than 50%.
Time Frame: Up to 3 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Number analyzed (Participants) | 19 | 0
Participants | 4 |

6. Other Pre Specified Outcome: Antiviral Effects (if Any in Those With HBV or HCV Associated HCC)
Time Frame: Up to 3 years
Population: Due to funding limitations, this outcome was not assessed.
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Drug Exposure, as Assessed by Steady State PK
Description: Associations between drug exposure and response/survival and toxicity by quartiles of drug exposure.
Time Frame: Up to 3 years
Population: Due to funding issues, data were not completed.
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Phase 1: Cycle 1 Day 15, Day 1 of Each Cycle After Cycle 1, Cycle 3 Day 1 (for phase 1 only), and to the End of Treatment. Phase II: From start of treatment until end of treatment.
Arm/Group | Treatment (Tivozanib 1mg) | Treatment (Tivozanib 1.5mg)
All-Cause Mortality (participants affected / at risk) | 18/24 | 3/3
Serious Adverse Events (participants affected / at risk) | 15/24 | 3/3
Other Adverse Events (participants affected / at risk) | 24/24 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tivozanib 1mg) (N=24) | Treatment (Tivozanib 1.5mg) (N=3)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tivozanib 1mg) (N=24) | Treatment (Tivozanib 1.5mg) (N=3)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (27) | 2 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 2 (2)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (23) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (12) | 1 (4)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (17) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 19 (45) | 2 (3)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 5 (5) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Perichondritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (7) | 2 (2)
Ammonia increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 5 (8) | 2 (2)
Blood bilirubin decreased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 6 (14) | 3 (6)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Lipase increased (Investigations) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (4) | 3 (8)
Platelet count decreased (Investigations) | 4 (5) | 2 (3)
Urine viscosity increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 8 (10) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 15 (28) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (7) | 3 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 10 (12) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 4 (5) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 2 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 1 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT01835223/Prot_SAP_000.pdf